CLINICAL TRIAL: NCT01729169
Title: Diagnosing Cardiac Sarcoidosis Using FDG PET: Optimization
Brief Title: Cardiac Sarcoidosis: FDG PET vs. Ga-DOTANOC PET
Status: Completed | Type: Observational
Sponsor: Lars Christian Gormsen (Other)
Responsible Party: Sponsor-Investigator, Lars Christian Gormsen, Consultant, MD PhD, Aarhus University Hospital
Organization: University of Aarhus (Other)
Other Study IDs: SarcoidosisPET
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Sarcoidosis; Cardiac Sarcoidosis
Keywords: Sarcoidosis; Cardiac sarcoidosis; 18-FDG PET; 68Ga-DOTANOC PET
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sarcoidosis patients: Patients with biopsy proven sarcoidosis suspected of having cardiac sarcoidosis

SUMMARY:
Diagnosing cardiac sarcoidosis has always been challenging: No single imaging modality has proved effective and cardiac biopsies have a very low sensitivity. 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) PET preceded by at least 12 hours of fasting has previously been demonstrated to have reasonable accuracy, however, in some patients physiological FDG uptake in the cardiac region hampers correct identification of sarcoid granulomas. Gallium Ga 68-DOTANOC is a conjugate of the somatostatin analogue Nal3-octreotide (NOC) and gallium Ga 68-labeled 1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetraacetic acid (DOTA). We aim to study whether 68Ga-DOTANOC has superior sensitivity and accuracy than 18-FDG PET in diagnosing cardiac sarcoidosis. In addition, we aim to compare 18-FDG PET preceded by 12 hours fasting with 18-FDG PET during somatostatin blockade of insulin mediated cardiac glucose uptake.

DETAILED DESCRIPTION:
Intervention:

* Study A: Subjects with biopsy proven sarcoidosis suspected of cardiac involvement (prone to arrhythmias, cardiac failure, unexplained dyspnea) are studied twice: 1) 18-FDG PET preceded by 12 hours fasting and 2) 18-FDG PET performed during a 2 hour somatostatin blockade (300 microgram/hour)/Heparin infusion.
* Study B: Subjects with biopsy proven sarcoidosis suspected of cardiac involvement are studied twice: 1) 18-FDG PET preceded by 12 hours fasting and 2) 68Ga-DOTANOC PET preceded by at least 6 hours fasting.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven sarcoidosis
* Suspected cardiac sarcoidosis

Exclusion Criteria:

* Ischemic heart disease
* Diabetes
* Cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy proven sarcoidosis suspected of having cardiac sarcoidosis
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Cardiac sarcoidosis - Sensitivity | 01/01/2015
  Ability to correctly identify patients with cardiac sarcoidosis

SECONDARY OUTCOMES:
Myocardial cardiac glucose uptake assessed by Cardiac SUV | 01/01/2015
  Semiquantitative assessment of myocardial glucose uptake, the Standardized Uptake Value (SUV). Expressed in g/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Gormsen LC, Haraldsen A, Kramer S, Dias AH, Kim WY, Borghammer P. A dual tracer (68)Ga-DOTANOC PET/CT and (18)F-FDG PET/CT pilot study for detection of cardiac sarcoidosis. EJNMMI Res. 2016 Dec;6(1):52. doi: 10.1186/s13550-016-0207-6. Epub 2016 Jun 17. PMID 27316444